CLINICAL TRIAL: NCT00057473
Title: A Phase II Study of Carboplatin Plus Irinotecan Versus Irinotecan in Children With Refractory Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA124-002
Record Dates: First submitted 2003-04-02; First posted 2003-04-03 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Neoplasms
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Neoplasms | interventions — Carboplatin; Irinotecan

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: carboplatin + irinotecan
- Arm B (Active Comparator)
  Interventions: Drug: irinotecan

INTERVENTIONS:
Drug: carboplatin + irinotecan — Solution, IV, Carbopaltin AUC 4 mg/ml.min every 21 days; irinotecan 12 mg/m2/day x 10 days , Minimum of two cycles of chemotherapy projected to be up to 6.
  Other Names: Paraplatin
  Arms: Arm A
Drug: irinotecan — Solution, IV, irinotecan 12 mg/m2/day x 10 days, minimum of two cycles of chemotherapy projected to be up to 6.
  Arms: Arm B

SUMMARY:
This clinical research study is being conducted to investigate the effectiveness of combining carboplatin and irinotecan, versus irinotecan alone, in treating children who have refractory solid tumors.

ELIGIBILITY:
* children 1-21 years of age
* confirmed diagnosis of measurable solid tumor, including brain tumor, which has progressed on or after standard therapy, or for which no effective standard therapy is known
* at least 4 weeks since last dose of immunotherapy, radiotherapy, or chemotherapy
* no more than 3 prior chemotherapies
* no symptomatic brain metastases

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2003-02; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
estimate response rate

SECONDARY OUTCOMES:
evaluate safety

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution, Orlando, Florida
  - Local Institution, Houston, Texas